CLINICAL TRIAL: NCT01102270
Title: A Double-Blind Randomized Physiological Study Examining the Effects of Eszopiclone on the Arousal Threshold and Obstructive Sleep Apnea Severity
Brief Title: The Effect of Eszopiclone on the Arousal Threshold in Sleep Apnea Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Atul Malhotra, MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2008P000818; 1P01HL095491-01 (NIH)
Record Dates: First submitted 2010-04-02; First posted 2010-04-13 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Arousal threshold; Sedative medication; upper airway
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Eszopiclone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eszopiclone (Active Comparator): Eszopiclone 3mg prior to sleep (1 night)
  Interventions: Drug: Eszopiclone
- Sugar Pill (Placebo Comparator): Sugar Pill (placebo) prior to sleep (1 night)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — 3mg tablet once prior to sleep
  Other Names: Lunesta
  Arms: Eszopiclone
Drug: Placebo — 1 placebo capsule prior to sleep
  Other Names: sugar pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to find out whether taking eszopiclone (Lunesta) changes the breathing effort required to briefly wake people with obstructive sleep apnea from sleep (respiratory arousal threshold). We would like to see if taking eszopiclone can reduce the severity of obstructive sleep apnea in some people (those that have a low respiratory arousal threshold; i.e. wake up easily to respiratory stimuli).

DETAILED DESCRIPTION:
Obstructive sleep apnea is an exceedingly common disease with major neurocognitive and cardiovascular consequences. The current primary treatment e.g. Continuous positive airway pressure (CPAP) is effective but poorly tolerated by many patients particularly those with mild-moderate disease. Secondary treatments such as oral appliances to advance the mandible or surgical procedures to enlarge the airway are commonly appealing to the patient. However, these approaches have only modest success in reducing apnea frequency to an acceptable level. Thus, finding tolerable and effective therapy for sleep apnea remains an important objective.

The causes of sleep apnea vary between patients. Targeted therapy according to the underlying causes of sleep apnea in individual patients is likely to be most effective. However, current therapeutic options for sleep apnea are quite limited. The purpose of this physiological research study is to determine if taking eszopiclone (Lunesta)changes the breathing effort required to briefly wake people with obstructive sleep apnea from sleep (the arousal threshold) and if administration of the sedative medication eszopiclone (Lunesta) to certain sleep apnea patients (those with a low arousal threshold ie wake up easily) would be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* Untreated obstructive sleep apnea

Exclusion Criteria:

* Nadir SaO2 <70% on a baseline PSG
* Medications known to affect either sleep, breathing or muscle activity
* Major co-morbidities apart from sleep apnea
* Allergy to lidocaine, oxymetazoline HCl, or eszopiclone
* Women who are pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Division of Sleep Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
published

REFERENCES:
- [Result] Eckert DJ, Owens RL, Kehlmann GB, Wellman A, Rahangdale S, Yim-Yeh S, White DP, Malhotra A. Eszopiclone increases the respiratory arousal threshold and lowers the apnoea/hypopnoea index in obstructive sleep apnoea patients with a low arousal threshold. Clin Sci (Lond). 2011 Jun;120(12):505-14. doi: 10.1042/CS20100588. PMID 21269278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects recruited 2008-2010 from clinics and ads
Groups:
- Eszopiclone First, Then Sugar Pill: Eszopiclone : 3mg tablet once prior to sleep followed by sugar pill (placebo) 1 week later
- Sugar Pill First, Then Eszopiclone: Placebo : 1 placebo capsule prior to sleep then 3mg eszopiclone 1 week later
Period: Overall Study
Arm/Group | Eszopiclone First, Then Sugar Pill | Sugar Pill First, Then Eszopiclone
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: although 28 were screened, only 17 were randomized since 11 did not qualify for the randomization portion of the study
Groups:
- All Study Participants: all study participants who received all interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Secondary Outcome: Arousal Threshold
Description: quantified using an epiglottic pressure transducer in CmH2O
Time Frame: 8 hour In-Laboratory Polysomnogram (PSG)
Measure: Median (Inter-Quartile Range); unit: cmH2O
Groups:
- Eszopiclone: Eszopiclone : 3mg tablet once prior to sleep
- Sugar Pill: Placebo : 1 placebo capsule prior to sleep
Arm/Group | Eszopiclone | Sugar Pill
Number analyzed (Participants) | 17 | 17
cmH2O | -18 [-22.1 to -15.1] | -14 [-19.9 to 10.9]

2. Secondary Outcome: Nadir Overnight Oxygen Saturation
Description: Nadir overnight oxygen saturation (%)
Time Frame: 8 hour In-Laboratory Polysomnogram (PSG)
Measure: Mean (Standard Error); unit: % oxygen saturation
Arm/Group | Eszopiclone | Sugar Pill
Number analyzed (Participants) | 17 | 17
% oxygen saturation | 80 (1) | 80 (1)

3. Primary Outcome: Apnea Hypopnea Index
Description: number of respiratory events per hour of sleep Respiratory events last for at least 10 seconds and are associated with a decrease in blood oxygenation or a cortical arosual from sleep. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and > 30/h = severe
Time Frame: 8 hour In-Laboratory Polysomnogram (PSG)
Measure: Mean (Standard Error); unit: events per hour of sleep
Arm/Group | Eszopiclone | Sugar Pill
Number analyzed (Participants) | 17 | 17
events per hour of sleep | 24 (4) | 31 (5)

4. Secondary Outcome: Sleep Duration
Description: total sleep duration
Time Frame: 8 hour In-Laboratory Polysomnogram (PSG)
Measure: Mean (Standard Error); unit: hours of sleep
Arm/Group | Eszopiclone | Sugar Pill
Number analyzed (Participants) | 17 | 17
hours of sleep | 6.8 (0.2) | 5.4 (0.4)

ADVERSE EVENTS:
Time Frame: Overnight study and the following morning
Arm/Group | Eszopiclone | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
We excluded patients with blood arterial oxygen saturations <70% as we wanted to avoid any potential risks associated with this group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No